CLINICAL TRIAL: NCT02264782
Title: PreView: The Preventive Video Education in Waiting Rooms Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 14988; NCI-2017-00456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14988 (Other: UCSF Medical Center-Mount Zion); R01CA158027 (NIH)
Record Dates: First submitted 2014-10-06; First posted 2014-10-15 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Health Status Unknown

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group I (PreView) (Experimental): Patients complete PreView, the Video Doctor plus Provider Alert, over 45 minutes on an iPad in the waiting room before a doctor visit.
  Interventions: Other: Computer-Assisted Intervention; Other: Questionnaire Administration
- Group II (educational video) (Active Comparator): Patients watch a video about healthy lifestyles including information about exercise and healthy eating over 45 minutes on an iPad in the waiting room before a doctor visit.
  Interventions: Other: Computer-Assisted Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Computer-Assisted Intervention — Complete PreView
  Arms: Group I (PreView)
Other: Computer-Assisted Intervention — Watch an educational video
  Arms: Group II (educational video)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well PreView, preventive video education, works in increasing rates of breast, cervical and colorectal cancer screening, improving participants' stage of change with respect to age appropriate cancer screening and increasing patient-provider discussions about prostate cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the extent to which PreView increases the likelihood that primary care patient participants will receive mammograms, pap tests, colon cancer tests or prostate specific antigen (PSA) testing discussions with primary care physicians compared with participants who receive usual care.

II. To determine the extent that PreView increases participants' readiness to be screened for breast cancer, cervical cancer or colorectal cancer (CRC) compared with usual care.

III. To determine the extent that PreView increases the likelihood that PSA testing will be discussed in primary care physician visits compared with usual care.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients complete PreView, the Video Doctor plus Provider Alert, over 45 minutes on an iPad in the waiting room before a doctor visit.

GROUP II: Patients watch a video about healthy lifestyles including information about exercise and healthy eating over 45 minutes on an iPad in the waiting room before a doctor visit.

ELIGIBILITY:
Inclusion Criteria:

* Without a history of cancer

Exclusion Criteria:

* With a history of cancer (for whom subsequent procedures would be surveillance and not screening)
* Individuals who do not speak English or Spanish (except for the testimonials)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2013-07; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Changing participants' readiness to be screened for breast, cervical and colorectal cancer | Up to 3 hours from pre-visit to post-visit interview.
  To determine the extent to which PreView increases the likelihood that primary care patient participants will receive mammograms, Pap tests, colon cancer tests or PSA testing discussions with primary care physicians compared with participants who receive usual care
Increasing physician-patient discussions about PSA screening measured by chart review | Baseline up to 14 months
  To determine the extent that PreView increases participants' readiness to be screened for breast cancer, cervical cancer or CRC compared with usual care.
Increasing rates of breast, cervical and colorectal cancer screening | From Baseline up to 14 months
  To determine the extent that PreView increases the likelihood that PSA testing will be discussed in primary care physician visits compared with usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Walsh, Principal Investigator — UCSF Medical Center-Mount Zion
Locations (2):
- United States (2):
  - John Muir Medical Center-Concord Campus, Concord, California
  - UCSF Medical Center-Mount Zion, San Francisco, California

REFERENCES:
- [Derived] Walsh J, Potter M, Salazar R, Ozer E, Gildengorin G, Dass N, Green L. PreView: a Randomized Trial of a Multi-site Intervention in Diverse Primary Care to Increase Rates of Age-Appropriate Cancer Screening. J Gen Intern Med. 2020 Feb;35(2):449-456. doi: 10.1007/s11606-019-05438-0. Epub 2019 Nov 14. PMID 31728894